CLINICAL TRIAL: NCT04877860
Title: Effectiveness of an E-Health System Integrated in a Physical Recovery Program for the Treatment of Pain in the Oncological Population. PaiNEd Study.
Brief Title: Pain Treatment in a Breast Cancer Population. PaiNEd Study.
Acronym: PaiNEd
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Carolina Fernández Lao, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI-0171-2020
Record Dates: First submitted 2021-03-18; First posted 2021-05-07 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
Keywords: E-health; exercise; telehealth; telerehabilitation; pain management; cancer
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Agnosia; Neoplasms | interventions — Exercise Therapy; Musculoskeletal Manipulations; Control Groups

STUDY DESIGN:
Intervention Model Description: Experimental design with two intervention groups and a control group. Effectiveness study.
  Intervention group 1: multimodal rehabilitation program + PNE Intervention group 2: multimodal rehabilitation program + traditional biomedical information Control group: Patient waiting list.
Who Masked: Participant, Care Provider
Masking Description: Participants who meet the inclusion criteria will be randomized into each of the groups using a random number generation program (EPIDAT 4.2, junta de Galicia). The sequence will be placed in an opaque envelope closed by a member outside the investigation and will be opened once the baseline assessment is completed, so the assessment staff will be masked for the randomization of the participants, thus reducing the risk of bias during the evaluation. The blinding of evaluators will be guaranteed by the fact that some members of the group are specialized in the treatment of cancer patients and others in their evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multimodal rehabilitation program + PNE (Therapeutic exercise, manual therapy and PNE) (Experimental): Physical recovery program (multimodal) with a duration of 8 weeks. Three weekly sessions on alternate days lasting 60 minutes each one. 4 individual manual therapy sessions (1 session every 2 weeks). Access to the PaiNEd system.
  Interventions: Other: Multimodal rehabilitation program + PNE (Therapeutic exercise, manual therapy and PNE)
- Multimodal rehabilitation program + traditional biomedical information (Active Comparator): Physical recovery program (multimodal) with a duration of 8 weeks. Three weekly sessions on alternate days lasting 60 minutes each one. 4 individual manual therapy sessions (1 session every 2 weeks). Dossier with traditional biomedical recommendations on the management of pain and disability.
  Interventions: Other: Multimodal rehabilitation program + traditional biomedical information
- Control group (Active Comparator): Information dossier with recommendations on pain control and dysfunction improvement.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Multimodal rehabilitation program + PNE (Therapeutic exercise, manual therapy and PNE) — The sessions will consist of therapeutic exercise in groups: a) warm-up (10 minutes aerobic exercise), b) active mobilizations (cervical / shoulder) c) strength exercises of the cervical and shoulder muscles + general conditioning d) active postural control e) stretching and relaxation exercises.
  4 sessions of myofascial induction.
  Finally, patients will have access to the PaiNEd system before the start of the program (to prepare them for treatment sessions) and during the development of the treatment program in which they will introduce their pain levels and their characteristics and also receive a series of educational advice and recommendations for its improvement.
  Arms: Multimodal rehabilitation program + PNE (Therapeutic exercise, manual therapy and PNE)
Other: Multimodal rehabilitation program + traditional biomedical information — The sessions will consist of therapeutic exercise in groups: a) warm-up (10 minutes aerobic exercise), b) active mobilizations (cervical / shoulder) c) strength exercises of the cervical and shoulder muscles + general conditioning d) active postural control e) stretching and relaxation exercises.
  4 sessions of myofascial induction.
  Patients will receive a dossier with traditional biomedical recommendations on pain management and disability associated with the side effects of cancer treatment.
  Arms: Multimodal rehabilitation program + traditional biomedical information
Other: Control group — Waiting list of patients who have agreed to participate in the study. They will receive an information dossier with recommendations on pain control and improvement of dysfunction (similar to what was worked on in the experimental group). These recommendations will be distributed at the beginning of the study (initial assessment) and they will be summoned at 8 weeks for the next collection of variables. All patients will be invited to participate in the experimental phase at the end of the control phase.
  Arms: Control group

SUMMARY:
The objectives of this study are: 1) To design and implement the PaiNEd system for the evaluation and treatment based on Pain Neuroscience Education (PNE) in cancer survivors with sequelae derived from medical treatments; 2) Study the effectiveness of the PaiNEd system integrated in a multimodal physical recovery program compared to traditional biomedical information.

This project aims to first carry out the design and implementation of an e-health system for the evaluation and treatment of pain. A randomized controlled experimental study will be carried out in which 72 breast cancer survivors will be recruited and randomly assigned to three study groups.

DETAILED DESCRIPTION:
People who have suffered cancer often do not find an adequate therapeutic response for the sequelae derived from its treatments. The objectives of this study are: 1) To design and implement the PaiNEd system for the evaluation and treatment based on Pain Neuroscience Education (PNE) in cancer survivors with sequelae derived from medical treatments; 2) Study the effectiveness of the PaiNEd system integrated in a multimodal physical recovery program compared to traditional biomedical information. In this regard, there is a shortage of proposals for certain subgroups of patients who demand special attention. This project aims to first carry out the design and implementation of an e-health system for the evaluation and treatment of pain. A randomized controlled experimental study will be carried out in which 72 breast cancer survivors will be recruited and randomly assigned to the three study groups: a) physical recovery program + access to the PaiNEd system; b) physical recovery program + traditional biomedical recommendations; c) control group. The evaluation will be carried out at baseline (at the beginning of the study), at 8 weeks (time of completion of the intervention) and at 6 months of follow-up of the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects over 18 years of age.
2. Having undergone surgery and finished adjuvant treatment (radiotherapy and / or chemotherapy) six months or two years ago.
3. Not having active cancer.
4. Having pain in the regions related to the tumor area (cervical and / or brachial and / or shoulder), pain ≥ 4 (VAS 0 to 10) for> 4 weeks
5. Present musculoskeletal or functional alterations in the previous regions.

Exclusion Criteria:

1. Identification by the research team of physical or mental impossibility to carry out the tests of the study.
2. Suffering from chronic pain or having suffered a previous trauma to the spine, head, temporomandibular joint or upper extremities.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Pain on the Visual Analogue scale and Brief Pain Inventory at 2 and 6 months. | Baseline, 2 and 6 months.
  The Visual Analogue Scale is used to assess the intensity of spontaneous neck, temporomandibular and shoulder pain. The VAS is a 100 mm line anchored with a '0' at one end representing no pain and '100' at the other end representing the worst pain imaginable.

SECONDARY OUTCOMES:
Changes from baseline in Pain Catastrophizing Scale at 2 and 6 months. | Baseline, 2 and 6 months.
  Used to assess catastrophic thinking related to pain. Pain catastrophizing scale is a 13-item self-reported questionnaire.
  Patients rate how frequent they experience each of 13 items or types of pain experience. It uses a 5-point Likert scale, from 0 (mild symptoms) to 4 (worst symptoms). The total score is derived from the sum of the individual scores for the 13 items. The higher the total score, the more the patient exhibits pain catastrophizing characteristics.
Changes from baseline in Central Sensitization Inventory (CSI) at 2 and 6 months. | Baseline, 2 and 6 months.
  Used to assess if participants have symptoms that may be related to central sensitisation.
  The Central Sensitization Inventory (CSI) is composed of two different parts. The first one consists of 25 statements, each answer is scored: 0 Never, 1 Rarely, 2 Sometimes, 3 Often, and 4 Always. So that, at most we will be able to obtain a score of 100 and a minimum of 0. The second part is a survey in which patients explain if they have been diagnosed of specific disorders. Higher CSI scores mean greater symptoms of central sensitization. If patients obtain a score greater than or equal to 40, we will consider that they have sufficient psychometrics to be correlated with central sensitization syndromes
Changes from baseline in Kinesiophobia on the Tampa Scale for Kinesiophobia (TSK-11) at 2 and 6 months. | Baseline, 2 and 6 months.
  Kinesiophobia will be measured by an 11-item version of the Tampa Scale for Kinesiophobia (TSK-11). Each item has 4 response options, "strongly disagree" scores 1 point, and "strongly agree" scores 4 points. The maximum possible score is 44 points and the minimum is 11 points. Greater scores mean strong fear of movement.
Changes from baseline in Active shoulder and cervical spine on goniometry at 2 and 6 months. | Baseline, 2 and 6 months.
  A plastic universal goniometer with two adjustable overlapping arms is used to objectively measure the active range of motion of the shoulder joint.
  An inclinometer device is used to objectively measure the active range of motion of the cervical joints.
Changes from baseline in Quality of life on The European Organization for Research and Treatment of Cancer Breast Cancer-Specific Quality of Life Questionnaire at 2 and 6 months. | Baseline, 2 and 6 months.
  This questionnaire is a breast cancer module of the The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire that contains 23 items rated on a four-point scale ranging from 1 (not at all) to 4 (very much). The items assess the side effects of therapy, arm symptoms, breast symptoms, body image, and sexual function. Additionally, there are single items assessing sexual enjoyment, anxiety caused by hair loss, and future outlook. The scores range between 0-100 points. For scales evaluating function, a higher score represents a higher level of functioning. For scales evaluating symptoms, a higher score indicates more severe symptoms.
Changes from baseline in Functional capacity on the The Six-Minute Walk Test at 2 and 6 months. | Baseline, 2 and 6 months.
  The Six-Minute Walk Test determines the maximum distance (meters) that a person can walk in 6 minutes. The participants are instructed to set their own pace, to "walk as far as they can in 6 minutes", and to volitionally increase or decrease the speed during the test. Standardized phrases of encouragement are given.
Changes from baseline in Isometric handgrip strength on Hand-held Dynamometry at 2 and 6 months. | Baseline, 2 and 6 months.
  Using manual isometric dynamometry with adjustable grip in a standing position with elbow in complete extension. The test is performed 3 times per hand (alternating both hands), with a 1-minute rest between trials. The average score for each hand is registered.
Changes from baseline in Strength endurance deep cervical musculature on cranio-cervical flexion test at 2 and 6 months. | Baseline, 2 and 6 months.
  This test measures the strength of the deep flexor muscles of the neck. It consists of placing the patient in supine position with the spine fully supported on the stretcher and asking him to first, to do a flexion of the upper cervical spine and to simultaneously flex the lower cervical spine. The time that the patient is able to maintain the position without loosing the initial distance that separated him from the stretcher is counted.
Changes from baseline in Body composition by using electrical bioimpedance analysis at 2 and 6 months. | Baseline, 2 and 6 months.
  The electrical impedance analysis is used for estimating body composition, in particular body fat and muscle mass.
Changes from baseline in stress and inflammatory responses at 2 and 6 months. | Baseline, 2 and 6 months.
  Salivary Cortisol, Interleukin-6 and C-reactive protein biomarkers are analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Fernández Lao, PhD, Study Director — Health Sciences Faculty, University of Granada
Locations (1):
- Health Sciences Faculty, University of Granada, Granada, Spain

REFERENCES:
- [Derived] Fernandez-Gualda MA, Ariza-Vega P, Lozano-Lozano M, Cantarero-Villanueva I, Martin-Martin L, Castro-Martin E, Arroyo-Morales M, Tovar-Martin I, Lopez-Garzon M, Postigo-Martin P, Gonzalez-Santos A, Artacho-Cordon F, Ortiz-Comino L, Galiano-Castillo N, Fernandez-Lao C. Persistent pain management in an oncology population through pain neuroscience education, a multimodal program: PaiNEd randomized clinical trial protocol. PLoS One. 2023 Aug 15;18(8):e0290096. doi: 10.1371/journal.pone.0290096. eCollection 2023. PMID 37582097